CLINICAL TRIAL: NCT03664102
Title: Comparison of Automated Fastener Device Versus Manually Tied Knot in Minimally-invasive Isolated Aortic Valve Replacement Surgery
Brief Title: Automated Fastener Device Versus Manually Tied Knot in MiAVR
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier La Chartreuse (Other)
Responsible Party: Principal Investigator, MORGANT Marie-Catherine, Principal investigator, Centre Hospitalier La Chartreuse
Other Study IDs: CCVT-MORGANT 082018
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Heart Valve Diseases
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sutures with hand-tied knots: Minimally-invasive isolated aortic valve replacement with Sutures were secured with hand-tied knots
- Sutures with automated fastener device (Cor-Knot): Minimally-invasive isolated aortic valve replacement with Sutures were secured with automated fastener device (Cor-Knot)
  Interventions: Device: Cor Knot

INTERVENTIONS:
Device: Cor Knot — Heart valve replacement with or without the use of automated fastener device Cor Knot
  Groups: Sutures with automated fastener device (Cor-Knot)

SUMMARY:
The aim of the investigator's study was to evaluate the efficacy and the safety of the Cor-Knot device in isolated aortic valve replacement (AVR) by right anterior minithoracotomy (RAMT).

Four hundred and forty patients were operated for AVR by RAMT. Of these patients, 221 underwent isolated AVR surgery with stented prosthesis. Sutures were secured using the Cor-Knot titanium fastener in 63 patients and knots were hand-tied in 158.

The aortic cross-clamping and cardiopulmonary bypass times were significantly decreased in the AT group compared with the MT group. Clinical outcomes were similar in the two groups, whether in the analysis of non-matched or matched groups. There was no difference in 30 day-mortality and the stroke and TIA rates were comparable The automated Cor-Knot fastener is an easy-to-use, time-saving device which does not increase perioperative morbi-mortality in patients undergoing AVR by right anterior minithoracotomy.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* Elective patient
* Isolated aortic valve replacement with stented prosthesis
* Minimally-invasive approach (right anterior minithoracotomy)

Exclusion Criteria:

* Associated procedure
* Aortic valve replacement with sutureless or rapid valve deployment prosthesis
* Active endocarditis
* Prior cardiac surgery

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient operated on an Isolated aortic valve replacement with stented prosthesis by Minimally-invasive approach (right anterior minithoracotomy)
Sampling Method: Non-Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2009-09-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-06 (Actual)

PRIMARY OUTCOMES:
Cardiac surgery times | peroperative data
  Aortic cross-clamping and cardiopulmonary bypass times

SECONDARY OUTCOMES:
Morbimortality | Perioperative (30 days) and 24 months follow up
  Morbidity (Stroke, pacemaker implantation, aortic regurgitation) Death Valve-related reoperation

IPD SHARING:
Plan to Share IPD: No
Trial on medical records only. No specific regulatory authorization required. The trial has already been recorded as Professionnal evaluation practices.